CLINICAL TRIAL: NCT05954104
Title: Evaluation of the Effect of Topical Calcipotriol Versus Platelet-Rich Plasma Versus Combined of Both on Serum Adiponectin Level in Alopecia Areata
Brief Title: Evaluation of the Effect of Topical Calcipotriol Versus Platelet-Rich Plasma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Faten Othman
Record Dates: First submitted 2023-06-23; First posted 2023-07-20 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata | interventions — calcipotriene

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Active Comparator): About 20 patients suffering from Alopecia areata , they will receive topical vit D3 analogue (calcipotriol) 0.005% twice daily for 3 months with follow up
  Interventions: Drug: Calcipotriol
- Group B (Active Comparator): About 20 patients suffering from Alopecia areata , they will be injected by PRP intra lesional for 3 consecutive sessions 4weeks apart.
  Interventions: Drug: Calcipotriol
- Group C (Active Comparator): About 20 patients suffering from Alopecia areata they will receive combined therapy ( PRP and topical vit D3 analogue).
  Interventions: Drug: Calcipotriol
- Group D (Active Comparator): About 20 of Healthy control group .
  Interventions: Drug: Calcipotriol

INTERVENTIONS:
Drug: Calcipotriol — To evaluate the efficacy of Calcipotriol on Alopecia Areata.
  Other Names: Platelet Rich Plasma

SUMMARY:
Alopecia areata (AA) is a common, immune-mediated non scarring alopecia and can be associated with severe psychological consequences . Alopecia Areata affects 2% of the global population. Alopecia Areata prevalence is lower in adults than children, is increasing over time, and significantly differs by region.

Its etiology is unknown but it was hypothesized to be an autoimmune disease mediated by T-lymphocytes. It has been suggested that inflammatory T cells induce growth arrest in hair bulbs in the anagen phase of the hair cycle . Cytotoxic T cells secrete tumor necrosis factor, granzymes, and Fas ligand which trigger apoptosis in affected hair follicle and disrupt hair growth

DETAILED DESCRIPTION:
Clinically, Alopecia Areata presents as a well-circumscribed patch of sudden hair loss. It affects any hair bearing area. The most common affected site is the scalp .

Dermoscopy is a highly valuable tool in diagnosis and follow-up of Alopecia Areata. The most common trichoscopic features of Alopecia Areata are yellow dots, micro exclamation mark hairs, tapered hairs, black dots, broken hairs, and regrowing upright or regrowing coiled hairs .

The diagnosis of alopecia areata is commonly established based on clinical appearance, In cases of ambiguity, trichoscopy may be useful to avoid invasive procedures such as biopsy.

Treatment of alopecia areata is dependent on age of patient as well as the extent and duration of scalp involvement. Treatments include steroids, topical immunotherapy, topical minoxidil, anthralin, and immunosuppressants. Each case must be dealt with on a customized individual basis.

Platelets rich plasma (PRP) is an autologous preparation of platelets in concentrated plasma. Injection of PRP improves cutaneous ischemic conditions, increases vascular structures around hair follicles and induces the proliferation of dermal papilla cells by up regulating fibroblast growth factor 7 (FGF-7) .Anagen-associated angiogenesis has been suggested as one of the important factors in active hair growth, due to the secretion of vascular endothelial growth factor by the keratinocytes of the outer root sheath and fibroblasts of the dermal papilla .

Topical calcipotriol is a vitamin D analogue that regulates keratinocytes proliferation and differentiation. It can induce hair regrowth in Alopecia Areata lesions by regulation of the differentiation of B cells, T cells, dendritic cells, and Toll-like receptor expression. There are few reports evaluating the effect of calcipotriol in Alopecia Areata .

Patients with Alopecia Areata are characterized by an abnormal serum level of adipokines, particularly adiponectin and resistin. Adiponectin may be considered as a marker of severity of hair loss in alopecia areata. Impaired secretion of specific adipokines may play an important and complex role in the pathogenesis of Alopecia Areata and its continuity

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-severe alopecia areata , a severity of alopecia tool (SALT) score up to 2 with less than 50% of scalp involvement.
* No restriction of age , race, nor occupation

Exclusion Criteria:

1. Pregnant and lactating women, immunocompromised patients.
2. Patients having active scalp inflammation.
3. Patients who received systemic treatment for Alopecia Areata in the last 3 months or applied any topical or intradermal treatments in the last 4 weeks .

Ages: 5 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Efficacy of topical calcipotriol and platelet Rich Plasma in Alopecia Areata treatment | from baseline to 3 months
  Evaluating the patients suffering from Alopecia Areata clinically, with Severity of Alopecia Tool (SALT) score. As score of 0 means no hair loss, while a SALT score of 100 is complete hair loss. and this evaluation will be done by trichoscopy

SECONDARY OUTCOMES:
serum adiponectin level. | from baseline to 3 months
  Compare the effect of topical calcipotriol, PRP, and combination of both on serum adiponectin level.by doing the ELISA test for Alopecia Areata patients before treatment and 3 months after treatment
serum Adiponectin level in Alopecia Areata | from baseline to 3 months
  Compare serum adiponectin level in Alopecia Areata patients with its serum level in healthy control group.by doing the ELISA test for Alopecia Areata patients before treatment and for healthy control group.

CONTACTS AND LOCATIONS:
Overall Officials: Moustafa Adam, Professor, Study Chair — Department of dermatology , Venerolgy and Andrology Faculty of Medicine Aswan university
Locations (1):
- Faculty of Dentistary - Aswan University, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No